CLINICAL TRIAL: NCT01511016
Title: The Effect of Leptin Therapy on Abnormal Lipid Kinetics in Subjects With HIV Lipodystrophy Syndrome
Brief Title: Leptin for Abnormal Lipid Kinetics in HIV Lipodystrophy Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Ashok Balasubramanyam, Professor of Medicine, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-13372
Record Dates: First submitted 2012-01-11; First posted 2012-01-18 (Estimated); Results first posted 2016-01-27 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2015-12

CONDITIONS: HIV Lipodystrophy
Keywords: lipid kinetics; fat oxidation
MeSH Terms: interventions — metreleptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- human recombinant leptin (metreleptin) (Experimental): Each subject received 0.02 mg leptin / kg body weight daily by subcutaneous injection for two months, followed by 0.04 mg leptin / kg for two more months.
  Interventions: Drug: Human recombinant leptin ("metreleptin")
- Placebo injection (Placebo Comparator): Each subject received placebo at a dose of 0.02 mg / kg body weight daily by subcutaneous injection for two months, followed by a dose of 0.04 mg / kg for two more months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human recombinant leptin ("metreleptin") — Metreleptin was administered at a dose of 0.02 mg / kg body weight for two months, followed by a dose of 0.04 mg / kg for two more months.
  Other Names: metreleptin
  Arms: human recombinant leptin (metreleptin)
Drug: Placebo — Placebo was administered at a dose of 0.02 mg / kg body weight daily by subcutaneous injection for two months, followed by 0.04 mg / kg for two more months.
  Arms: Placebo injection

SUMMARY:
"HIV lipodystrophy syndrome" (HLS) is characterized by loss of fat in the arms and legs, with increase in fat in the abdomen, and abnormal blood lipid levels. Persons with HLS have high risk for cardiovascular disease and diabetes mellitus and the metabolic syndrome. The investigators have previously shown that the abnormal lipid levels and lipodystrophy in HLS are associated with defective regulation of lipid metabolic rates, specifically, accelerated lipolysis (breakdown of stored fats), and decreased fat oxidation (utilization of fats for energy). Patients with HLS also have low levels of the hormone leptin. The investigators hypothesize that treatment of these patients with leptin will improve fat oxidation and may slow the rate of lipolysis. Hence, the investigators propose to study the effect of leptin therapy on lipid metabolic rates and lipid and glucose levels in adults with HLS. The investigators will use state of the art stable isotope tracer techniques and gas chromatography mass spectrometry (GCMS) to measure lipolysis, fat oxidation, and fat re-esterification in adipose tissues and liver.

DETAILED DESCRIPTION:
The HIV lipodystrophy syndrome (HLS) is characterized by peripheral fat wasting and central obesity, and hyperlipidemia (mainly hypertriglyceridemia), which results in insulin resistance. HLS patients are at high risk for cardiovascular disease, diabetes mellitus and the metabolic syndrome.

The investigators have previously shown that the alterations in lipid metabolism in the so-called mixed form of HLS are due to dysregulation of lipid kinetics at two levels. First, there appears to be an acceleration in lipid kinetics, with higher total and net lipolysis despite higher intra-adipocyte re-esterification. However, the percentage of fatty acid flux being oxidized remains the same, leading to increased hepatic recycling of fatty acids to triglycerides (TG), and export of TG-rich VLDL into the circulation. Second, there is reduced clearance of chylomicron and VLDL-TG from the plasma, resulting in the striking hypertriglyceridemia associated with this syndrome. The investigators propose that these alterations in lipid kinetics account for the phenotypic changes characteristic of this syndrome: increased lipolysis would facilitate peripheral lipoatrophy, increased intra-adipocyte re-esterification (if selective in intrabdominal depots) would contribute to the central obesity, and increased hepatic re-esterification together with impaired VLDL- and chylomicron-TG clearance would lead to hypertriglyceridemia.

Rational treatment of HLS should be targeted at these fundamental kinetic defects. Leptin is in many ways an ideal agent, since it increases fat oxidation, and shifts the ratio of utilization of free fatty acids derived from lipolysis towards oxidation and away from re-esterification, and decreases plasma triglyceride levels. HLS patients with lipoatrophy have low circulating levels of leptin. Moreover, leptin has been shown to be effective in correcting similar defects in fat redistribution and circulating lipids in non-HIV forms of lipodystrophy. Hence, the investigators propose to study (using a blinded, placebo-controlled, dose escalating design) the effect of leptin therapy on lipid kinetics and fat distribution in adult subjects with the lipoatrophic and mixed (peripheral lipoatrophy and central adiposity) forms of HLS. The investigators will use state of the art stable isotope tracer techniques and gas chromatography mass spectrometry (GCMS) to measure whole body lipolysis, lipid oxidation, lipid re-esterification and hepatic lipid recycling.

ELIGIBILITY:
Inclusion Criteria:

* predominantly lipoatrophic or mixed phenotype of HIV-lipodystrophy (based on self-observation and evaluation by a study physician utilizing a visual scale;
* AM fasting leptin < 4.0 ng/ml
* hypertriglyceridemia (fasting serum TG 250-1000 mg /dl).
* normal biochemistry (except altered lipid and glucose profile). Patients with the American Diabetes Association diagnostic criteria for diabetes were included provided the HbA1c level was <7.5% and they received no anti-diabetic medications for at least 3 months.
* well-controlled HIV infection status evidenced by viral RNA titers <400 copies/ml, on stable HAART.

Exclusion Criteria:

* acute or chronic illnesses.
* use of antidiabetic medications in the previous 3 months, or of lipid-lowering drugs in the previous 6 weeks are also exclusion criteria. Other drugs excluded are growth hormone (if used without evidence of growth hormone deficiency), Megace and testosterone (if used without evidence of hypogonadism).

Ages: 18 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2003-02; Primary Completion 2011-06 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ashok Balasubramanyam, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- [Result] Sekhar RV, Jahoor F, Iyer D, Guthikonda A, Paranilam J, Elhaj F, Coraza I, Balasubramanyam A. Leptin replacement therapy does not improve the abnormal lipid kinetics of hypoleptinemic patients with HIV-associated lipodystrophy syndrome. Metabolism. 2012 Oct;61(10):1395-403. doi: 10.1016/j.metabol.2012.03.013. Epub 2012 Apr 28. PMID 22542724

RESULTS

PARTICIPANT FLOW:
Recruitment Details: HIV-positive subjects meeting the entry criteria were recruited from March, 2003 until November, 2010 from the clinics of Harris County Hospital District, and Legacy Community Health Center, Houston.
Pre-assignment Details: If a potential study subject was already taking a lipid lowering medication at the time of screening but was otherwise eligible for the study, he/she was invited to stop the medication for 6 weeks, at the end of which the fasting triglyceride level was re-measured to gauge eligibility.
Groups:
- Placebo Injection: Each subject will receive placebo at a dose of 0.02 mg / kg body weight daily by subcutaneous injection for two months, followed by a dose of 0.04 mg / kg for two more months.
  Placebo : Placebo will administered at a dose of 0.02 mg / kg body weight daily by subcutaneous injection for two months, followed by 0.04 mg / kg for two more months.
- Human Recombinant Leptin (Metreleptin): Each subject will receive 0.02 mg leptin / kg body weight daily by subcutaneous injection for two months, followed by 0.04 mg leptin / kg for two more months.
  Human recombinant leptin ("metreleptin") : Metreleptin will be administered at a dose of 0.02 mg / kg body weight for two months, followed by a dose of 0.04 mg / kg for two more months.
Period: Overall Study
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Started | 8 | 9
Completed | 6 | 7
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin) | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 9 | 17
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.1 (6.8) | 44.9 (7.8) | 46.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 8 | 9 | 17
Region of Enrollment [Number; unit: participants]
  United States | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Rate of Total Lipolysis
Description: Rate of total lipolysis was measured in plasma samples by mass spectrometry following stable isotope infusions of labeled glycerol and palmitate
Time Frame: 4 months after treatment
Population: Subjects in each group were analyzed and compared after 4 months of treatment.
Measure: Mean (Standard Error); unit: mmol FFA/kg/h
Groups:
- Placebo Injection: Each subject received placebo at a dose of 0.02 mg / kg body weight daily by subcutaneous injection for two months, followed by a dose of 0.04 mg / kg for two more months.
  Placebo : Placebo was administered at a dose of 0.02 mg / kg body weight daily by subcutaneous injection for two months, followed by 0.04 mg / kg for two more months.
- Human Recombinant Leptin (Metreleptin): Each subject received 0.02 mg leptin / kg body weight daily by subcutaneous injection for two months, followed by 0.04 mg leptin / kg for two more months.
  Human recombinant leptin ("metreleptin") : Metreleptin was administered at a dose of 0.02 mg / kg body weight for two months, followed by a dose of 0.04 mg / kg for two more months.
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Number analyzed (Participants) | 8 | 9
mmol FFA/kg/h | 0.649 (0.073) | 0.767 (0.137)

2. Secondary Outcome: Rates of Fatty Acid Oxidation
Description: Rates of fatty acid oxidation were measured in breath samples following stable isotope infusions of 13C-labeled palmitate.
Time Frame: 4 months after treatment
Population: Number of subjects in each group remaining at the end of 4 months of treatment.
Measure: Mean (Standard Error); unit: mmol FFA/kg/h
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Number analyzed (Participants) | 6 | 8
mmol FFA/kg/h | 0.239 (0.023) | 0.214 (0.040)

3. Secondary Outcome: Fasting Plasma Non-HDL-C
Description: Fasting plasma non-HDL-cholesterol was calculated from measured total cholesterol and HDL cholesterol.
Time Frame: 4 months after treatment.
Population: Number of subjects in each group remaining after 4 months of treatment.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Number analyzed (Participants) | 6 | 8
mg/dL | 136 (9) | 127 (7)

4. Secondary Outcome: Glucose Levels After Glucose Challenge
Description: An oral glucose tolerance test was performed. This is not PD/PK in the sense that we are not studying the distribution or clearance of a drug. Rather, we are performing a standard clinical test of glucose tolerance. i.e., a test for diabetes and pre-diabetes. Although multiple time points are used in this test, the outcome is a single value, either a blood glucose level after 2 hours or an area-under-the-curve. In this study we are reporting the area-under-the-curve.
Time Frame: 4 months after treatment.
Population: Number of subjects remaining after 4 months of treatment.
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Number analyzed (Participants) | 4 | 5
mg/dL | 6268 (434) | 6647 (514)

5. Secondary Outcome: Insulin Levels After Oral Glucose Challenge.
Description: An oral glucose tolerance test was performed to measure endogenous insulin response. This is not PD/PK in the sense that we are not studying the distribution or clearance of a drug. Rather, we are performing a clinical test of endogenous insulin response to glucose i.e., an endocrine test. Although multiple time points are used in this test, the outcome is a single value, i.e., an area-under-the-curve for insulin.
Time Frame: 4 months after treatment.
Population: Number of subjects remaining after 4 months of treatment.
Measure: Mean (Standard Error); unit: microU/mL
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Number analyzed (Participants) | 4 | 5
microU/mL | 1580 (954) | 2868 (890)

6. Primary Outcome: Rate of Net Lipolysis
Description: Rate of net lipolysis was measured in plasma samples by mass spectrometry following stable isotope infusions of labeled glycerol and palmitate
Time Frame: 4 months after treatment
Population: Subjects in each group were analyzed and compared after 4 months of treatment
Measure: Mean (Standard Error); unit: mmol FFA/kg/h
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Number analyzed (Participants) | 8 | 9
mmol FFA/kg/h | 0.386 (.074) | 0.508 (.106)

ADVERSE EVENTS:
Time Frame: The duration of the study for each subject was 4 months. However, due to slow recruitment the entire study took place over approximately 4 years; therefore the average duration of subject follow-up for Adverse Events was approximately 2 years
Arm/Group | Placebo Injection | Human Recombinant Leptin (Metreleptin)
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Injection (N=8) | Human Recombinant Leptin (Metreleptin) (N=9)
Hyperthyroidism (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Weight loss (Metabolism and nutrition disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
1. Relatively small sample size.
2. Early drop-out of 3 subjects (2 in placebo arm, 2 in metreleptin arm).
3. Possible confounders in phenotypic hetereogeneity of HIV lipodystrophy, and differences in antiretroviral drugs.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No